CLINICAL TRIAL: NCT04648384
Title: Association of Whey Protein and Casein in the Same Proportions of Human Breast Milk Promoted Similar Branched-chain Amino Acids Profile and Reduced Delayed Muscle Soreness in Physically Active Man
Brief Title: Acute Whey Protein And Casein Supplementation: Effect On Protein Metabolism After Resistance Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government); Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government); Instituto Colombiano para el Desarrollo de la Ciencia y la Tecnología (COLCIENCIAS) (Other Government)
Responsible Party: Principal Investigator, Ellen Cristini de Freitas, Principal Investigator, University of Sao Paulo
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: Protein Supplementation
Record Dates: First submitted 2020-11-09; First posted 2020-12-01 (Actual); Last update posted 2020-12-02 (Actual); Status verified 2020-11

CONDITIONS: Sports Nutrition; Protein Supplementation
MeSH Terms: interventions — Resistance Training

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Protein Supplementation and Resistance exercise (Experimental): Protein supplementation composed of 20 gram of whey protein or casein in different proportions (80:20) and fasting state 10 sets of 10 reps at 85% of 1 Maximum repetition
  Interventions: Dietary Supplement: Blend Protein Supplementation; Other: Resistance Exercise
- Placebo Supplementation (Placebo Comparator): Placebo supplementation composed of 20 gram of Maltodextrin and fasting state 10 sets of 10 reps at 85% of 1 Maximum repetition
  Interventions: Dietary Supplement: Placebo Supplementation; Other: Resistance Exercise
- Resistance Training (Experimental): Resistance Exercise will be performed before supplementation and is composed by 10 sets of 10 repetitions at 85% of 1 Maximum repetition in leg press exercise.
  Interventions: Other: Resistance Exercise

INTERVENTIONS:
Dietary Supplement: Blend Protein Supplementation — Protein supplementation using 20 grams of whey protein or casein mix. Acute Resistance training, 10 sets of 10 reps at 85% of 1Maximum repetition
  Other Names: Resistance Training
  Arms: Protein Supplementation and Resistance exercise
Dietary Supplement: Placebo Supplementation — Placebo supplementation using 20 grams of Maltodextrin. Acute Resistance training, 10 sets of 10 reps at 85% of 1Maximum repetition
  Other Names: Resistance Training
  Arms: Placebo Supplementation
Other: Resistance Exercise — 10 sets of 10 repetitions at 85% of 1 Maximum repetition in leg press exercise

SUMMARY:
The proteins of human breast milk are the most important endocrine signaling system that promotes neonatal growth by increasing the release of insulin, insulin-like growth factor-1 (IGF-1), and the leucine-mediated mammalian target of rapamycin complex 1- (mTORC1) signaling of pancreatic β-cells. Remarkably, the branched-chain amino acids (BCAAs) leucine, isoleucine, and valine are involved in the growth-promoting effects of milk, protein biosynthesis, and metabolism because they physiologically stimulate insulin secretion The present study sought to investigate the effects of the combination of whey protein and casein in the ratio of 80:20 ("whey protein: casein" or "casein: whey protein") as breast milk proportion on the peak and the period of the permanence of branched-chain amino acids in the blood circulation, final metabolites of protein metabolism and delayed onset muscle soreness (DOMS) after a single bout of fasting or a resistance exercise session.

DETAILED DESCRIPTION:
The present study investigated the effects of the association of WP and casein in the ratio of 80:20, a similar ratio of human breast milk, on blood branched-chain amino acids (BCAAs) profile by HPLC technique, markers of protein metabolism (creatinine, urea, and urine nitrogen) and delayed onset muscle soreness (DOMS) after a single bout of resistance exercise. A double-blind, crossover and acute study was conducted with ten men (age 29 ± 8 y; BMI: 25.4 ± 2.9 Kg/m2; 77 ± 12 kg; 1.74 ± 0.09 m) that were randomly assigned to five supplementation treatments: WP - whey protein; CAS - casein; WP/CAS - 80% WP/20% CAS; CAS/WP - 80% CAS/ 20% WP; PLA - placebo. Participants were submitted to the following evaluations: performance sessions, blood collection for each session for the BCAAs profile determination, two food records, 3-days assessment of DOMS (24h, 48h, 72h) after each treatment.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* practice resistance training at least 3x a week

Exclusion Criteria:

* Smokers
* Muscle injures
* cardiovascular diseases
* Diabetes mellitus
* Lactose intolerance

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2016-03-20 (Actual); Primary Completion 2019-07-20 (Actual); Study Completion 2019-10-20 (Actual)

PRIMARY OUTCOMES:
Change from baseline in plasma amino acids concentration | 5 weeks
  Blood sample collected for analysis of BCAA concentration after blend protein or placebo supplementation expressed in (µmol/L)
Change from baseline in 1RM test | 5 weeks
  Change of training load using RPE, time and load expressed in (a.u)
Change in protein metabolism | 5 weeks
  Change in nitrogen excretion, and nitrogen balance after protein supplementation expressed in (g/24 hours)
Changes from baseline in macronutrient intake | 5 weeks
  Change of macronutrient intake were calculated pre and post treatment expressed in (g/24 hours)
Change in delayed onset muscle soreness | 5 weeks
  Change from baseline the delayed onset muscle soreness pre, post, 24 hours, 48 hours and 72 hours after treatment expressed in (a.u)

CONTACTS AND LOCATIONS:
Locations (1):
- University of São Paulo, School of Physical Education and Sports of Ribeirão Preto., Ribeirão Preto, São Paulo, Brazil

REFERENCES:
- [Derived] Martinez Galan BS, Giolo De Carvalho F, Carvalho SCS, Cunha Brandao CF, Morhy Terrazas SI, Abud GF, Meirelles MSS, Sakagute S, Ueta Ortiz G, Marchini JS, Aristizabal JC, Cristini de Freitas E. Casein and Whey Protein in the Breast Milk Ratio: Could It Promote Protein Metabolism Enhancement in Physically Active Adults? Nutrients. 2021 Jun 23;13(7):2153. doi: 10.3390/nu13072153. PMID 34201617